CLINICAL TRIAL: NCT03748368
Title: Computer-based Tutorial as Supportive Means to Enhance Quality and Efficiency of the Informed Consent Process for Cataract Surgery in Turkish or Serbian Speaking Patients
Brief Title: Computer-based Tutorial for the Informed Consent Process for Cataract Surgery in Turkish or Serbian Speaking Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Prim. Prof. Dr. Oliver Findl, MBA (Other)
Responsible Party: Sponsor-Investigator, Prim. Prof. Dr. Oliver Findl, MBA, Principal Investigator, Vienna Institute for Research in Ocular Surgery
Organization: Vienna Institute for Research in Ocular Surgery (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: CatInfo SK/TK
Record Dates: First submitted 2018-11-19; First posted 2018-11-20 (Actual); Last update posted 2019-10-02 (Actual); Status verified 2019-10

CONDITIONS: Cataract
Keywords: Cataract surgery; Informed Consent Process
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cataract presentation (Active Comparator): Cataract presentation prior to surgery
  Interventions: Other: Cataract presentation
- Placebo presentation (Placebo Comparator): Placebo presentation prior to surgery
  Interventions: Other: Placebo presentation

INTERVENTIONS:
Other: Cataract presentation — Presentation about cataract surgery
  Arms: Cataract presentation
Other: Placebo presentation — Presentation about the history of the hospital
  Arms: Placebo presentation

SUMMARY:
Investigate if a computer-based tutorial enhances the quality and efficiency of the informed consent process for cataract surgery in Turkish or Serbian speaking patients.

DETAILED DESCRIPTION:
Informing the patient and obtaining informed consent is one of the major duties physicians have to perform before beginning a medical treatment. However, patients often experience the informed consent taking as not satisfying. In the past, several approaches were used to try to improve the informed consent taking, such as printed information sheets and multimedia tools.

A novel concept introduced several years ago is to use a multimedia tool including a so-called traffic light system. The patient sees and hears information concerning cataract surgery on a touch screen and after each short chapter a traffic light is shown on the touch screen. At this point the patient has to decide, whether everything is clear and he wants to continue (green light), if he has further questions for the ophthalmologist (yellow light), or if he wants to repeat the chapter (red light). The patient's feedback for each chapter is then printed and guides the ophthalmologist during the face to face interview. This approach is called "CatInfo tool".

The German version of the CatInfo tool has been developed and evaluated in a previous study. In short, the CatInfo tool was developed as a multidisciplinary project including patients, graphic designers and ophthalmologists. The first version of the tool was evaluated in patient focus-groups. Afterwards, an evaluation study including 60 patients was performed. Main outcome was the following: patients who used the CatInfo tool were significantly better informed than patients only having a face to face interview with an ophthalmologist and the feedback concerning the CatInfo tool was good. Meanwhile the German version of the CatInfo tool is part of our daily routine and thousands of patients profited from the CatInfo tool consent always additional to the face to face interview with an ophthalmologist. However, some patients are not able to use the CatInfo tool. One reason is that they are not literate in German. Aim of this study is to translate and evaluate a Serbian and Turkish version of the CatInfo tool to allow better access.

ELIGIBILITY:
Inclusion Criteria:

* Cataract
* Age 21 and older
* First eye to be operated
* No previous ophthalmic surgery
* Written informed consent to participation in the study

Exclusion Criteria:

* Not literate in Serbian (Serbian group) / Turkish (Turkish group) or German (both groups)
* Visual acuity of less than 6/60 in the worse eye
* Severe hearing loss
* Inability to use touch screen device (e.g. severe tremor, etc.)
* Pregnancy - for women in the reproductive age a pregnancy test is required

Ages: 21 Years to 105 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2020-05-01 (Estimated); Study Completion 2020-07-01 (Estimated)

PRIMARY OUTCOMES:
Number of correctly answered questions between study group and control group | 12 months
  Patients are asked to complete a multiple choice questionnaire concerning cataract surgery. Correctly answered questions will be summated. The scale ranges from a minimum of 0 points to a maximum of 19 points. The more points the better the patients knowledge about cataract

SECONDARY OUTCOMES:
Usability of the touchscreen device | 12 months
  By using an audiovisual analogue scale ranging from 0 (worst usability) to 10 (best usability) patients will be asked about their impression concerning usability of the CatInfo tool

CONTACTS AND LOCATIONS:
Locations (1):
- Vienna Institute for Research in Ocular Surgery (VIROS), Vienna, Austria

IPD SHARING:
Plan to Share IPD: Undecided